CLINICAL TRIAL: NCT06260566
Title: A Phase 1 Trial of Tolerability of Enteral N-Acetylcysteine in Infants
Brief Title: Tolerability of Enteral NAC in Infants
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sanjiv Harpavat (Other)
Collaborators: Baylor College of Medicine (Other)
Responsible Party: Sponsor-Investigator, Sanjiv Harpavat, Associate Professor, Baylor College of Medicine
Organization: Baylor College of Medicine (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: H-52570
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Biliary Atresia
Keywords: Biliary Atresia; N-Acetylcysteine; glutathione; bile flow; serum bilirubin; serum bile acids; cholestasis
MeSH Terms: conditions — Biliary Atresia; Cholestasis | interventions — Acetylcysteine

STUDY DESIGN:
Intervention Model Description: The study consists of two parts:
  * Administering applesauce alone (lead-in): In study days 1-2, infants will receive one infant spoon (approximately ½ teaspoon) of plain applesauce by mouth twice a day. If the infant tolerates 3-4 of 4 total doses without emesis, the infant will progress to the final two days of the study.
  * Administering applesauce plus NAC (for infants who tolerate applesauce in study days 1-2): In study days 3-4, infants will receive an individualized dose of powdered oral NAC mixed into one infant spoon of applesauce by mouth twice a day for a maximum of four doses of NAC medication.
Masking Description: N/A. No Masking
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Infants with Biliary Atresia (Experimental): * Administering applesauce alone
  * Administering applesauce plus NAC (for infants who tolerate applesauce alone)
  Interventions: Drug: N-Acetylcysteine

INTERVENTIONS:
Drug: N-Acetylcysteine — This is a phase 1 study of tolerance of a novel delivery method of oral NAC medication in infants with biliary atresia. The study consists of two parts:
  * Administering applesauce alone (lead-in): In study days 1-2, infants will receive one infant spoon (approximately ½ teaspoon) of plain applesauce by mouth twice a day. If the infant tolerates 3-4 of 4 total doses without emesis, the infant will progress to the final two days of the study.
  * Administering applesauce plus NAC (for infants who tolerate applesauce in study days 1-2): In study days 3-4, infants will receive an individualized dose of powdered oral NAC mixed into one infant spoon of applesauce by mouth twice a day for a maximum of four doses of NAC medication. 4 doses will be trialed: 150 mg/kg/day, 240 mg/kg/day, 330 mg/kg/day, and 420 mg/kg/day using BOIN study design for dose escalation.
  Other Names: NAC

SUMMARY:
Biliary atresia (BA) is a neonatal liver disease characterized by impaired bile flow and is the most common indication for pediatric liver transplantation. BA can be treated with the Kasai portoenterostomy (KP), a procedure that attempts to restore bile flow and slow disease progression. However, success of the KP procedure is quite variable, and lack of adjuvant medical therapies following KP is a major gap in pediatric hepatology.

This study begins to explore oral N-acetylcysteine (NAC) as a potential medical therapy in BA by determining whether an oral formulation can be given to infants. The primary objective is to determine tolerability of the oral NAC formulation. The primary outcome is tolerating at least 3 out of 4 total doses without emesis. The Bayesian Optimal Interval Design (BOIN) trial design will be used to determine the maximum tolerated dose of oral NAC. Our secondary objective is to assess palatability of the oral NAC formulation by comparing facial expressions when taking oral NAC versus other medications commonly given to cholestatic infants.

DETAILED DESCRIPTION:
Biliary atresia (BA), a neonatal liver disease characterized by impaired bile flow, is the most common indication for pediatric liver transplantation. The only identified treatment option other than liver transplant is a Kasai portoenterostomy (KP). This surgical procedure directly connects the intestines to the liver in an attempt to restore bile flow. By restoring bile flow and decreasing bile retention, the KP's goal is to slow disease progression. Restored bile flow within the first 3-6 months post-operatively is associated with better clinical outcomes. Unfortunately the success of the procedure is quite variable with one-third of KPs never achieving sufficient bile flow to slow disease progression and the remaining one-third never achieving any bile flow. These patients go on to require liver transplantation with 60% of liver transplants in infants <1 year of age and 30% of all pediatric liver transplants being performed for BA. The lack of adjuvant medical therapies for KP is a major gap in the current field of pediatric hepatology.

NAC is an attractive potential therapy for BA, because NAC is the precursor for glutathione. Glutathione in turn addresses much of the problematic pathophysiology in biliary atresia including poor bile flow, oxidative damage, and inflammation. Preclinical studies have demonstrated that glutathione in the form of NAC therapy has been shown to improve liver histology in various rodent models of cholestasis and biliary atresia. In a recent study by Luo et al, rotavirus-induced mouse models of biliary atresia were injected with saline for placebo or 150 mg/kg/day NAC. The mice that received NAC demonstrated better weight gain, decreased hepatic injury, and improved survival when compared to mice that received saline. Liver biopsies demonstrate decreased inflammation, epithelial injury, and portal inflammation in the RRV-induced BA mice that received NAC (RRV+NAC; right two panels) when compared to RRV-induced BA mice that received placebo saline injections (RRV+PBS; middle two panels). These results support the notion that glutathione may reduce inflammation and fibrosis, perhaps by preventing oxidative damage caused by retained bile.

Luo et al also reported clinical data that demonstrated cholestatic infants with upregulation of genes related to regulating glutathione metabolism had improved survival rates at two years of age, lending further support to the hypothesis that glutathione can improve outcomes in cholestatic infants. There is a list of gene groups from livers of patients with biliary atresia at time of diagnosis that were discovered to be upregulated in patients that demonstrated improved survival with their native liver at two years of age. Notably genes for glutathione metabolism, glutathione biosynthesis, and glutathione conjugation were all upregulated in the patients with improved survival with their native liver. This suggests that increased glutathione is associated with improved survival in patients with BA.

An important advantage of NAC therapy is that it is been shown to be safe in both pre-term and term infants with other conditions such as increased risk for chorioamnionitis. Prolonged intravenous (IV) NAC therapy has also been demonstrated to be safe in infants with other liver conditions such as cholestasis secondary to total parental nutrition. Additionally, IV NAC was given to infants and children with non-acetaminophen induced liver failure in similar doses as proposed in this study and there was no significant difference in rates of adverse events between the treatment and control groups.

While NAC is a promising therapeutic agent post-KP that has been demonstrated to be safe in multiple previous studies, the only study to date investigating NAC in BA used an IV formulation (study performed at Texas Children's Hospital, data analysis in process). An IV formulation is the logical choice when infants are on bowel rest immediately post-KP and remain hospitalized with IV access. However, discharging a patient home with indwelling venous access poses a substantial infection risk with up to 30% of peripherally inserted central catheters having at least one complication. Transitioning to oral NAC prior to discharge home would allow for longer duration of therapy without the potential consequences of indwelling venous access, however oral NAC has a sulfuric, unpleasant taste.

To address the unpleasant taste of oral NAC, the investigators plan to utilize novel powdered NAC - which has a less sulfuric flavor and odor when compared to typical NAC solution - mixed into a small amount of applesauce just prior to oral administration. This method of medication administration is frequently utilized to give pancreatic enzymes to infants with cystic fibrosis as young as one week of age. Additionally, as the goal of this study is to determine if oral NAC can be safely administered to relatively well infants with BA that will be starting purees around 4-6 months of age, the risk of choking and aspiration should be no greater than baseline.

These infants will be captured for the 2-4 day study when admitted to the hospital for other indications such as fever, concern for cholangitis, or expedited liver transplantation evaluation. These hospitalizations are frequent, and infants typically are stable and do not require intensive care unit care. As infants with BA are typically initially very clinically stable with a slow decline in synthetic liver function and overall health during the first year of life, most infants eligible for study inclusion will be relatively healthy and eating by mouth at time of being approached for study inclusion. This will also eliminate any increased risk of choking or aspiration.

The ultimate goal of this trial is to demonstrate that infants with biliary atresia are able to tolerate oral NAC prior to proposing and conducting a prolonged efficacy trial of NAC in relatively well infants with BA in an ambulatory setting.

The investigators hypothesize that infants will tolerate this novel administration of oral NAC. To test this hypothesis, the investigators will perform a two-part study. In the first part, applesauce will be administered and its tolerability assessed. In the second part, only those infants who tolerated applesauce will receive up to four total doses of oral applesauce plus NAC medication over the course of two days. The primary outcome will be measured only in infants taking applesauce plus NAC and based on total number of doses without emesis (defined as forceful oral expulsion of any milk/formula, medication, or gastric content containing liquid). The secondary outcomes are infants' facial expressions when taking applesauce or applesauce plus NAC compared to their facial expression when taking other medications routinely given to cholestatic infants, such as ursodeoxycholic acid and fat-soluble vitamins. Other secondary outcomes are adverse events occurring during applesauce and applesauce plus NAC administration. This study employs the Bayesian Optimal Interval (BOIN) design, which was initially developed for phase 1 oncology trials and allows for a higher probability of identifying the maximum tolerated dose with a small sample size.

ELIGIBILITY:
Inclusion Criteria:

* 122-273 days of life at time of enrollment
* Confirmed diagnosis of biliary atresia based on intraoperative cholangiogram
* Able to tolerate oral nutrition and medications and not on continuous tube feeds
* Anticipated inpatient admission of at least 4 days
* Legal guardian(s) consent to study enrollment after understanding the risks and investigational nature of the study

Exclusion Criteria:

* Gestational age of <32 weeks at birth
* Inability or contraindication to taking oral nutrition
* Neonatal intensive care unit admission
* Short bowel, or other malabsorptive, syndrome
* Decompensated liver disease (INR > 1.3 despite vitamin K administration)
* Active respiratory infection
* Severe concurrent illnesses that would interfere with the conduct and/or results of the study
* Concurrent participation in another drug trial

Ages: 122 Days to 273 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
No emesis within 30 minutes of administration of at least 3 of 4 total doses of oral NAC | within 30 minutes
  No emesis with administration of at least 3 of 4 total doses of oral NAC

SECONDARY OUTCOMES:
Oral NAC palatability compared to clinically indicated medications using the facial expression scale | at the time of adminsitration
  Facial expression scale uses visual facial expressions scored 0-5 with higher scores indicating worse outcome
Oral NAC-specific adverse event evaluation | 28 days
  Adverse event severity grade scale scored 1 - 5 with 5 indicating worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Harpavat, M.D., PH.D., Principal Investigator — Baylor College of Medicine - Texas Children's Hospital

IPD SHARING:
Plan to Share IPD: No
IPD will not be available to other researchers.

REFERENCES:
- [Background] Squires RH, Ng V, Romero R, Ekong U, Hardikar W, Emre S, Mazariegos GV. Evaluation of the pediatric patient for liver transplantation: 2014 practice guideline by the American Association for the Study of Liver Diseases, American Society of Transplantation and the North American Society for Pediatric Gastroenterology, Hepatology and Nutrition. Hepatology. 2014 Jul;60(1):362-98. doi: 10.1002/hep.27191. No abstract available. PMID 24782219
- [Background] Bezerra JA, Wells RG, Mack CL, Karpen SJ, Hoofnagle JH, Doo E, Sokol RJ. Biliary Atresia: Clinical and Research Challenges for the Twenty-First Century. Hepatology. 2018 Sep;68(3):1163-1173. doi: 10.1002/hep.29905. PMID 29604222
- [Background] Shneider BL, Magee JC, Karpen SJ, Rand EB, Narkewicz MR, Bass LM, Schwarz K, Whitington PF, Bezerra JA, Kerkar N, Haber B, Rosenthal P, Turmelle YP, Molleston JP, Murray KF, Ng VL, Wang KS, Romero R, Squires RH, Arnon R, Sherker AH, Moore J, Ye W, Sokol RJ; Childhood Liver Disease Research Network (ChiLDReN). Total Serum Bilirubin within 3 Months of Hepatoportoenterostomy Predicts Short-Term Outcomes in Biliary Atresia. J Pediatr. 2016 Mar;170:211-7.e1-2. doi: 10.1016/j.jpeds.2015.11.058. Epub 2015 Dec 24. PMID 26725209
- [Background] Karrer FM, Price MR, Bensard DD, Sokol RJ, Narkewicz MR, Smith DJ, Lilly JR. Long-term results with the Kasai operation for biliary atresia. Arch Surg. 1996 May;131(5):493-6. doi: 10.1001/archsurg.1996.01430170039006. PMID 8624194
- [Background] Sundaram SS, Mack CL, Feldman AG, Sokol RJ. Biliary atresia: Indications and timing of liver transplantation and optimization of pretransplant care. Liver Transpl. 2017 Jan;23(1):96-109. doi: 10.1002/lt.24640. PMID 27650268
- [Background] Tessier MEM, Shneider BL, Brandt ML, Cerminara DN, Harpavat S. A phase 2 trial of N-Acetylcysteine in Biliary atresia after Kasai portoenterostomy. Contemp Clin Trials Commun. 2019 May 2;15:100370. doi: 10.1016/j.conctc.2019.100370. eCollection 2019 Sep. PMID 31193715
- [Background] Luo Z, Shivakumar P, Mourya R, Gutta S, Bezerra JA. Gene Expression Signatures Associated With Survival Times of Pediatric Patients With Biliary Atresia Identify Potential Therapeutic Agents. Gastroenterology. 2019 Oct;157(4):1138-1152.e14. doi: 10.1053/j.gastro.2019.06.017. Epub 2019 Jun 19. PMID 31228442
- [Background] Galicia-Moreno M, Favari L, Muriel P. Antifibrotic and antioxidant effects of N-acetylcysteine in an experimental cholestatic model. Eur J Gastroenterol Hepatol. 2012 Feb;24(2):179-85. doi: 10.1097/MEG.0b013e32834f3123. PMID 22241216
- [Background] Tahan G, Tarcin O, Tahan V, Eren F, Gedik N, Sahan E, Biberoglu N, Guzel S, Bozbas A, Tozun N, Yucel O. The effects of N-acetylcysteine on bile duct ligation-induced liver fibrosis in rats. Dig Dis Sci. 2007 Dec;52(12):3348-54. doi: 10.1007/s10620-006-9717-9. Epub 2007 Apr 12. PMID 17436097
- [Background] Galicia-Moreno M, Rodriguez-Rivera A, Reyes-Gordillo K, Segovia J, Shibayama M, Tsutsumi V, Vergara P, Moreno MG, Muriel P. N-acetylcysteine prevents carbon tetrachloride-induced liver cirrhosis: role of liver transforming growth factor-beta and oxidative stress. Eur J Gastroenterol Hepatol. 2009 Aug;21(8):908-14. doi: 10.1097/MEG.0b013e32831f1f3a. PMID 19398917
- [Background] Jenkins DD, Wiest DB, Mulvihill DM, Hlavacek AM, Majstoravich SJ, Brown TR, Taylor JJ, Buckley JR, Turner RP, Rollins LG, Bentzley JP, Hope KE, Barbour AB, Lowe DW, Martin RH, Chang EY. Fetal and Neonatal Effects of N-Acetylcysteine When Used for Neuroprotection in Maternal Chorioamnionitis. J Pediatr. 2016 Jan;168:67-76.e6. doi: 10.1016/j.jpeds.2015.09.076. Epub 2015 Nov 3. PMID 26545726
- [Background] Mager DR, Marcon M, Wales P, Pencharz PB. Use of N-acetyl cysteine for the treatment of parenteral nutrition-induced liver disease in children receiving home parenteral nutrition. J Pediatr Gastroenterol Nutr. 2008 Feb;46(2):220-3. doi: 10.1097/MPG.0b013e3180653ce6. No abstract available. PMID 18223385
- [Background] Kortsalioudaki C, Taylor RM, Cheeseman P, Bansal S, Mieli-Vergani G, Dhawan A. Safety and efficacy of N-acetylcysteine in children with non-acetaminophen-induced acute liver failure. Liver Transpl. 2008 Jan;14(1):25-30. doi: 10.1002/lt.21246. PMID 18161828
- [Background] Squires RH, Dhawan A, Alonso E, Narkewicz MR, Shneider BL, Rodriguez-Baez N, Olio DD, Karpen S, Bucuvalas J, Lobritto S, Rand E, Rosenthal P, Horslen S, Ng V, Subbarao G, Kerkar N, Rudnick D, Lopez MJ, Schwarz K, Romero R, Elisofon S, Doo E, Robuck PR, Lawlor S, Belle SH; Pediatric Acute Liver Failure Study Group. Intravenous N-acetylcysteine in pediatric patients with nonacetaminophen acute liver failure: a placebo-controlled clinical trial. Hepatology. 2013 Apr;57(4):1542-9. doi: 10.1002/hep.26001. Epub 2013 Feb 4. PMID 22886633
- [Background] Barrier A, Williams DJ, Connelly M, Creech CB. Frequency of peripherally inserted central catheter complications in children. Pediatr Infect Dis J. 2012 May;31(5):519-21. doi: 10.1097/INF.0b013e31824571b0. PMID 22189533
- [Background] Atkuri KR, Mantovani JJ, Herzenberg LA, Herzenberg LA. N-Acetylcysteine--a safe antidote for cysteine/glutathione deficiency. Curr Opin Pharmacol. 2007 Aug;7(4):355-9. doi: 10.1016/j.coph.2007.04.005. Epub 2007 Jun 29. PMID 17602868
- [Background] AbbVie Inc. "Creon (Pancrelipase) Delayed-Release Capsule: Official Website - Tips for Giving Enzymes to Your Baby." 2017, https://www.creon.com/infants/infantdosing. Accessed 2022.
- [Background] Yuan Y, Hess KR, Hilsenbeck SG, Gilbert MR. Bayesian Optimal Interval Design: A Simple and Well-Performing Design for Phase I Oncology Trials. Clin Cancer Res. 2016 Sep 1;22(17):4291-301. doi: 10.1158/1078-0432.CCR-16-0592. Epub 2016 Jul 12. PMID 27407096
- [Background] Smilkstein MJ, Knapp GL, Kulig KW, Rumack BH. Efficacy of oral N-acetylcysteine in the treatment of acetaminophen overdose. Analysis of the national multicenter study (1976 to 1985). N Engl J Med. 1988 Dec 15;319(24):1557-62. doi: 10.1056/NEJM198812153192401. PMID 3059186
- [Background] Rumack BH, Peterson RC, Koch GG, Amara IA. Acetaminophen overdose. 662 cases with evaluation of oral acetylcysteine treatment. Arch Intern Med. 1981 Feb 23;141(3 Spec No):380-5. doi: 10.1001/archinte.141.3.380. PMID 7469629
- [Background] Viscomi C, Burlina AB, Dweikat I, Savoiardo M, Lamperti C, Hildebrandt T, Tiranti V, Zeviani M. Combined treatment with oral metronidazole and N-acetylcysteine is effective in ethylmalonic encephalopathy. Nat Med. 2010 Aug;16(8):869-71. doi: 10.1038/nm.2188. Epub 2010 Jul 25. PMID 20657580
- [Background] Tirouvanziam R, Conrad CK, Bottiglieri T, Herzenberg LA, Moss RB, Herzenberg LA. High-dose oral N-acetylcysteine, a glutathione prodrug, modulates inflammation in cystic fibrosis. Proc Natl Acad Sci U S A. 2006 Mar 21;103(12):4628-33. doi: 10.1073/pnas.0511304103. Epub 2006 Mar 13. PMID 16537378
- [Background] Hardan AY, Fung LK, Libove RA, Obukhanych TV, Nair S, Herzenberg LA, Frazier TW, Tirouvanziam R. A randomized controlled pilot trial of oral N-acetylcysteine in children with autism. Biol Psychiatry. 2012 Jun 1;71(11):956-61. doi: 10.1016/j.biopsych.2012.01.014. Epub 2012 Feb 18. PMID 22342106
- [Background] Seattle Children's Hospital. "Medicine - Refusal to Take." 2022. https://www.seattlechildrens.org/conditions/a-z/medicine-refusal-to-take/. Accessed 2022.
- [Background] Acetylcysteine solution, USP10% and 20%teartop vials. labeling.pfizer.com. (n.d.). https://labeling.pfizer.com/ShowLabeling.aspx?id=4101
- [Background] Mullins ME, Schmidt RU Jr, Jang TB. What is the rate of adverse events with intravenous versus oral N-acetylcysteine in pediatric patients? Ann Emerg Med. 2004 Nov;44(5):547-8; author reply 548-9. doi: 10.1016/j.annemergmed.2004.03.051. No abstract available. PMID 15523751